CLINICAL TRIAL: NCT02326350
Title: ASpirin as a Treatment for ARDS (STAR): a Phase 2 Randomised Control Trial
Acronym: STAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Queen's University, Belfast (Other); Northern Ireland Clinical Trials Unit (Other)
Responsible Party: Principal Investigator, Professor Danny McAuley, Professor and consultant of Intensive Care Medicine, Belfast Health and Social Care Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14043DMcA-AS
Record Dates: First submitted 2014-12-16; First posted 2014-12-29 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress syndrome; Aspirin
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin 75mg (Experimental): Aspirin 75mg enterally once daily for a maximum of 14 days
  Interventions: Drug: Aspirin 75mg
- Placebo (Placebo Comparator): Lactose powder placebo enterally once daily for a maximum of 14 days
  Interventions: Drug: Lactose powder

INTERVENTIONS:
Drug: Aspirin 75mg — Active treatment
  Arms: Aspirin 75mg
Drug: Lactose powder — Placebo
  Arms: Placebo

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) causes the lungs to fail due to the collection of fluid in the lungs (pulmonary oedema). ARDS is common in severely ill patients in Intensive Care Units and is associated with a high mortality and a high morbidity in those who survive. There is a large economic burden with direct healthcare costs, but also indirectly due to the impact on the carer and patient through their inability to return to full time employment. There is little evidence for effective drug (pharmacological) treatment for ARDS. Blood cells called platelets have increasingly been recognized to play a key role in the development of ARDS. There is increasing information that aspirin, a drug which is widely used to treat heart disease, might be important in treating ARDS. We plan to test if aspirin will help in the treatment of ARDS. To do this we will divide patients suffering from ARDS into two groups, one of which will get aspirin and the other a harmless dummy (or placebo) tablet who will then be followed up to determine if lung function improves. If effective this may lead to further research to determine if aspirin is effective in patients with ARDS. This project will also provide new information about mechanisms in the development of ARDS leading, potentially, to other new treatments.

DETAILED DESCRIPTION:
The role of aspirin as a novel therapy for ARDS.

Aspirin inhibits cyclo-oxygenase enzymes, therefore preventing the formation of lipid mediators including thromboxane A2 (TxA2) and pro-inflammatory prostaglandins from arachidonic acid. TxA2 is required for platelet degranulation and aggregation. Production of pro-inflammatory prostaglandins from arachidonic acid is mediated by cyclo-oxygenase-2 (COX-2), an enzyme induced in inflammatory and endothelial cells by cytokines, growth factors and bacterial products including lipopolysaccharide (LPS). Prostaglandin E2 (PGE2) is a key downstream pro-inflammatory product of COX-2 activation. It can act in an auto and paracrine fashion on local inflammatory and parenchymal cells to increase intracellular cyclic adenosine mono-phosphate (cAMP), drive nuclear translocation of NFκB and thus the production of many pro-inflammatory cytokines, including TNFα and IL-8. Aspirin can also induce the production of a lipoxin (aspirin-triggered 15-epi-lipoxin A4, also known as ATL). Lipoxins are a group of anti-inflammatory eicosanoids derived from arachidonic acid which act via the lipoxin A4 receptor (LXA4R) on leucocytes to inhibit free-radical formation, and reduce activation of the proinflammatory transcription factors AP-1 and NFκB, all of which are implicated in the development of ARDS.

Hypothesis.

Treatment with aspirin is safe and improves important surrogate clinical outcomes in adult patients with ARDS.

Trial objectives.

To conduct a randomised, double-blind, allocation concealed, placebo-controlled phase 2 trial of aspirin as a treatment for ARDS.

To study the biological effects of aspirin on pulmonary and systemic inflammatory responses, epithelial and endothelial function and injury and lipid inflammatory mediators.

Population.

Patients will be prospectively screened daily. All patients with ARDS will be entered into a screening log. If the patient is not recruited the reason will be recorded, this will ensure the study can be reported in keeping with CONSORT guidelines (www.consort-statement.org). Routinely collected patient demographics will also be collected on these patients. This will allow comparison to identify that the study population is representative of the overall cohort of patients. We have an established and effective system in place to screen and identify patients with ARDS.

Informed consent procedure.

The study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki. The chief investigator (CI) is responsible for ensuring that informed consent for trial participation is given by each patient or a legal representative. An appropriately trained doctor or nurse may take consent. Appropriate signatures and dates must be obtained on the informed consent documentation prior to collection of trial data and administration of the trial drug. If no consent is given a patient cannot be randomised into the trial.

The incapacitating nature of the condition precludes obtaining prospective informed consent from participants. In this situation informed consent will be sought from a Personal Legal Representative or Professional Legal representative.

Personal legal representative consent.

Informed consent will be sought from the patient's personal legal representative (Per LR) who may be a relative, partner or close friend. The Per LR will be informed about the trial by the responsible clinician or a member of the research team and provided with a copy of the covering statement for the Per LR with an attached participant information sheet (PIS) and asked to give an opinion as to whether the patient would object to taking part in such medical research. If the Per LR decides that the patient would have no objection to participating in the trial they will be asked to sign two copies of the Per LR consent form which will then be countersigned by the person taking consent. The Per LR will retain one copy of the signed consent form. The second copy will be photocopied and the photocopy placed in the patients' medical records whilst the original will be retained in the trial site file.

Professional legal representative consent.

As the patient is unable to give informed consent and no Per LR is available, a doctor who is not connected with the conduct of the trial may act as a professional legal representative (Prof LR). The doctor will be informed about the trial by the responsible clinician or a member of the research team and given a copy of the PIS. If the doctor decides that the patient is suitable for entry into the trial they will be asked to sign two copies of the professional legal representative consent form. The doctor will retain one copy of the signed consent form. The second copy will be photocopied and the photocopy placed in the patient's medical records; the original will be retained in the trial site file.

Retrospective patient consent.

Patients will be informed of their participation in the trial by the responsible clinician or a member of the research team once they regain capacity to understand the details of the trial. The responsible clinician or a member of the research team will discuss the study with the patient and the patient will be given a copy of the PIS to keep. The patient will be asked for consent to participate in the trial and to sign two copies of the consent to continue form which will then be countersigned by the person taking consent. The patient will retain one copy of the signed consent form. The second copy will be photocopied and the photocopy placed in the patient's medical records whilst the original will be retained in the trial site file.

Where consent to continue is not obtained, consent from the legal representative will remain valid. If the patient refuses consent, permission to use data collected to that point and to access medical records for trial data will be requested from the patient.

Withdrawal of consent.

Patients may withdraw or be withdrawn (by Per LR or Prof LR) from the trial at any time without prejudice and consent will be requested to use the data collected to that point. If a patient or Per LR requests termination of the trial drug during the treatment period, the drug will be stopped but the patient will continue to be followed-up as part of the trial. If a patient or a Per LR withdraws consent during trial treatment, the trial drug will be stopped but permission will be sought to access medical records for data related to the trial. If a patient or Per LR wishes to withdraw from the trial after completion of trial treatment, permission to access medical records for trial data will be sought.

Randomisation.

Patients in the STAR study are eligible for co-enrolment in other non-CTIMP studies, this will be decided on a case by case basis.

Randomisation procedure.

The clinical trials pharmacist will be provided with a randomisation schedule which has been generated by the CTU. After informed consent, the researcher will contact the clinical trials pharmacist who will allocate the next sequential number as per the randomisation schedule. Randomisation will be stratified by vasopressor use. The clinical trials pharmacist will dispense the trial drugs. Study drug will be dispensed as per local pharmacy guidelines. Aspirin and placebo study drug will have an identical appearance. The researcher will then register the recruited patient with the CTU.

Study procedures for unblinding.

The investigator or treating physician may unblind a participant's treatment assignment in the case of an emergency, when knowledge of the study treatment is essential for the appropriate clinical management or welfare of the subject. Should a treating clinician require emergency unblinding, they should contact the clinical trials pharmacist at the Royal Victoria Hospital during working hours or if out of working hours the on call pharmacist for the Belfast Health and Social Care Trust for emergency unblinding. Following this and once the patient is stable, all reasonable efforts should then be made to contact the CI or co-Investigators who will be contactable via an emergency contact telephone number The date and reason for the unblinding must be recorded in the CRF.

Study drug

Treatment regimen.

Subjects will be randomised to receive aspirin 75mg capsule or a placebo capsule enterally for up to 14 days. Subjects will be randomised in a 1:1 ratio using blocks of variable size. The first dose of the study drug will ideally be administered within 4 hours of randomisation and subsequent doses will be as close to 10 am as possible starting on the following calendar day.

Study drug compliance.

Any omission of the study drug will be recorded in the CRF to monitor compliance.

Study drug accountability.

The clinical trials pharmacist will be responsible for maintaining records of the study drug dispensed to patients in ICU including dates, quantity, lot number and expiry date. Drug administration will be recorded on the patient's prescription chart.

Study drug return and destruction.

At the end of the treatment period any remaining unused drug will be returned to the hospital pharmacy. Destruction of trial medication will be in accordance with pharmacy department's standard operating procedures (SOPs) and hospital waste management policy. A record of destruction will be maintained.

Standardised management.

All patients will receive standardised management with regards to nutrition, antibiotic policy, fluid management and weaning. Patients will be managed using a standardised mechanical ventilation protocol aiming for tidal volumes of 6 ml/kg ideal body weight.

The influence of other treatments provided to critically ill patients will be minimised as the study will be undertaken in a single centre where standardised care is delivered based on evidence based local guidelines.

Data collection and recording.

All data for an individual patient will be collected by the CI or their delegated nominees and recorded in the CRF. CRFs are to be submitted to the CTU as per the CRF Submission Schedule.

Patient identification in the CRF will be through their unique Subject Number allocated at the time of randomisation and initials. Data will be collected from the time the patient is considered for entry into the trial through to their discharge from hospital.

Submitted data will be reviewed for completeness and entered onto a secure, backed-up custom database. Due care will be taken to ensure data safety and integrity, and compliance with the Data Protection Act 1998.

Data censorship will occur after 90 days post randomisation.

Training Issues.

To ensure accurate, complete and reliable data, the CTU will do the following:

* Be available for consultation with the trial personnel by mail, telephone and/or fax.
* Review and evaluate CRF data, detect errors in data collection and request data verification.

Data management.

Following the submission of CRFs to the CTU, the data will be processed as per the CTU SOPs. Data queries will be generated for site staff as required to clarify data or request missing information. The designated site staff will be required to respond to these queries within 2 weeks and send them back to the CTU after they have been reviewed and signed by the CI/delegated staff member. Any amended information will then be entered in the study database. A copy of the signed data query form should be retained with the CRF at the investigator site.

Data storage.

All essential documentation and trial records will be stored by the CI in conformance with the applicable regulatory requirements and access to stored information will be restricted to authorised personnel.

Statistical considerations.

Sample size.

The primary outcome measure will be the difference in OI between the aspirin and placebo treated groups at day 7. Based on our data from a recently completed clinical trial in ARDS, the mean (standard deviation; SD) OI at day 7 in patients with ARDS is 62 (51) cmH2O/kPa. A sample size of 56 subjects (28 in each group) will have 80% power at a two-tailed significance level of 0.05 to detect a clinically significant difference of 39 cmH2O/kPa in OI between groups. In a previous phase 2 study of similar size, we have found that an intervention can demonstrate a change in OI of a similar magnitude confirming a treatment effect of this size can be achieved.

Although we anticipate few withdrawals or loss to follow-up we have allowed for this in the sample size calculation. In our previous single centre study of simvastatin in ARDS there were no withdrawals. In a multi-centre UK study of pulmonary artery catheters in ICU patients (PAC-Man), no patients were lost to follow up, and only 3% withdrew consent after recovering competency. This is in keeping with our local data. Therefore a drop-out rate of 5% has been estimated and the study will require a total of 60 patients (30 in each group).

Statistical analysis.

For continuously distributed outcomes, differences between groups will be tested using independent samples t-tests and analysis of covariance with transformations of variables to normality if appropriate, or non-parametric equivalents. Chi-square tests (or Fisher's Exact tests) will be used for categorical variables. A secondary analysis excluding patients identified to have aspirin resistance will also be undertaken. The study will be analysed with an intention to treat so all randomised patients will be included in the analysis. A p value of 0.05 will be considered as significant.

Correlations between changes in the biological markers measured and physiological and clinical outcomes will be assessed by appropriate graphical and statistical methods including Pearson's (or Spearmans) correlation coefficient.

A single final analysis is planned at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving invasive mechanical ventilation.
2. ARDS as defined by the Berlin definition.

   * Onset within 1 week of identified insult.
   * Within the same 24 hours

     * Hypoxic respiratory failure (PaO2/ FiO2 ratio ≤ 40kPa on PEEP ≥ 5 cmH20),
     * Bilateral infiltrates on chest X-ray consistent with pulmonary oedema not explained by another pulmonary pathology,
     * No evidence of heart failure or volume overload

Exclusion Criteria:

1. More than 72 hours from the onset of ARDS.
2. Age < 16 years.
3. Patient is known to be pregnant.
4. Participation in a clinical trial of an investigational medicinal product within 30 days.
5. Current treatment with aspirin or within the past 4 weeks.
6. Platelet count < 50 x 109/l.
7. Haemophilia or other haemorrhagic disorder or concurrent therapeutic anticoagulant therapy.
8. History of aspirin sensitive asthma or nasal polyps associated with asthma.
9. Active or history of recurrent peptic ulcer and/ or gastric/ intestinal haemorrhage or other kinds of bleeding such as cerebrovascular haemorrhage.
10. Traumatic brain injury.
11. Active gout.
12. Currently receiving methotrexate.
13. Severe chronic liver disease with Child-Pugh score > 12.
14. Known hypersensitivity or previous adverse reaction to salicylic acid compounds or prostaglandin synthetase inhibitors.
15. Physician decision that aspirin is required for proven indication.
16. Contraindication to enteral drug administration, e.g. patients with mechanical bowel obstruction.
17. Treatment withdrawal imminent within 24 hours.
18. Consent declined.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-02-06 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
Oxygenation index (OI) | Day 7
  OI is a physiological index of the severity of ARDS and measures both impaired oxygenation and the amount of mechanical ventilation delivered.

SECONDARY OUTCOMES:
Oxygenation index | Days 4 and 14
Sequential organ failure assessment (SOFA) score | Days 4, 7 and 14
  SOFA score is a measure of organ failure
Respiratory compliance (Crs) | Days 4, 7 and 14
  Crs is a physiological measure of pulmonary function in ARDS
Partial pressure of arterial oxygen to the fraction of inspired oxygen ratio (P/F ratio) | Days 4, 7 and 14
  P/F ratio is a physiological measure of pulmonary function in ARDS
Safety and tolerability as assessed by the occurrence of serious adverse events and suspected unexpected serious adverse reactions | Up to 28 days after completion of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Danny F McAuley, Professor, Principal Investigator — Belfast Health and Social Care Trust

REFERENCES:
- [Derived] Toner P, Boyle AJ, McNamee JJ, Callaghan K, Nutt C, Johnston P, Trinder J, McFarland M, Verghis R, McAuley DF, O'Kane CM. Aspirin as a Treatment for ARDS: A Randomized, Placebo-Controlled Clinical Trial. Chest. 2022 May;161(5):1275-1284. doi: 10.1016/j.chest.2021.11.006. Epub 2021 Nov 14. PMID 34785236
- [Derived] Toner P, McAuley DF, Shyamsundar M. Aspirin as a potential treatment in sepsis or acute respiratory distress syndrome. Crit Care. 2015 Oct 23;19:374. doi: 10.1186/s13054-015-1091-6. PMID 26494395